CLINICAL TRIAL: NCT00782483
Title: Personalized Interactive Laser Therapy of Port Wine Stain - Study 2
Brief Title: Personalized Interactive Laser Therapy of Port Wine Stain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI moved out of state.
Sponsor: University of Arkansas (Other)
Collaborators: Arkansas Children's Hospital Research Institute (Other); Children's University Medical Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 104344; UAMS Sponsored
Record Dates: First submitted 2008-10-29; First posted 2008-10-31 (Estimated); Results first posted 2014-07-21 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-06

CONDITIONS: Port Wine Stain
Keywords: Diagnosis; Port Wine Stain; PWS
MeSH Terms: conditions — Port-Wine Stain; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: ThermoVision A20M Infrared Camera — FLIR Systems, Boston, MA. This is a non invasive passive thermal imaging device with less than minimal risk to subjects and staff.
Device: ScleroPLUS — Sclerolaser, Candela Corp., Wayland, MA. This laser is approved by the food and drug administration (FDA) for treating PWS lesions and will be used as labeled.
Device: 3D Digital Camera — 3dMD, Atlanta, GA. Approved by the food and drug administration (FDA) for imaging patients and will be used as labeled.

SUMMARY:
Lasers are being used to treat Port Wine Stains (PWS), but the laser doesn't always work. Only about 10% of PWS can be completely cleared. The research team believes that the investigators can improve the response of PWS to laser therapy by using a computer program that the principal investigator of this study (Dr. Shafirstein PhD) has developed. The purpose of this study is to test the validity of this computer program. Personalized Interactive Laser Therapy (PILT) could significantly improve clinical outcomes of laser treatment of PWS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with a PWS
* At least one visible PWS measuring greater than or equal to 15 mm in diameter.
* Information provided regarding alternative treatment methods, includig no treatment.
* Reading, understanding, and signing of an informed consent document.
* Children age 7 years or older has read, understood, and signed an assent document.
* Agreement to participate in the study.
* Agreement to return to at least 1 follow-up evaluation and treatment within 1 year after first treatment.
* Zubrod performance status of 0 or 1 at screening.

Exclusion Criteria:

* Inability or unwillingness of subject to participate in the study.
* Inability or unwillingness of one parent or legal guardian of the subject to sign written informed consent document.
* Subject can not return to at least 1 follow-up visit within 1 year, after the first treatment.

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2008-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gal Shafirstein, PhD, Principal Investigator — UAMS, ACH
Locations (1):
- Arkansas Children's Hospital, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Laser Therapy: Total number of participants
Period: Overall Study
Arm/Group | Laser Therapy
Started | 6 (6 subjects enrolled beginning on 04/27/2009 with last enrollment on 04/13/2010.)
Completed | 0
Not Completed | 6
Not completed — Early Termination of Protocol - PI Reloc | 6

BASELINE CHARACTERISTICS:
Groups:
- Overall: Overall Study Group
Arm/Group | Overall
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Average Laser Setting to be Used to Treat Port Wine Stains as Measured by Mathematical Calculations Based on Imaging and Temperature Analysis of Malformation.
Description: 6 subjects were enrolled but no data was ever collected due to early termination of the study due to the PI's relocation.
Time Frame: Three treatments up to one year, whichever is first
Population: 6 subjects were enrolled but no data was ever collected due to early termination of the study due to the PI's relocation.
Arm/Group | Laser Therapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Overall
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

LIMITATIONS AND CAVEATS:
PI relocated and protocol was terminated, and no subject returned for treatment under protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No